CLINICAL TRIAL: NCT03110315
Title: A Double-blind, Crossover, Placebo-controlled Study to Compare the Effects of Nighttime Administration of Suvorexant in Patients With Multiple Sclerosis Fatigue and Insomnia
Brief Title: A Study of Suvorexant in Patients With Multiple Sclerosis Fatigue and Insomnia
Acronym: DREAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Theodore R. Brown, MD MPH (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Theodore R. Brown, MD MPH, Principal Investigator, EvergreenHealth
Organization: EvergreenHealth (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TRB 2017.2
Record Dates: First submitted 2017-03-28; First posted 2017-04-12 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis; Fatigue; Insomnia
Keywords: Multiple Sclerosis; Fatigue; Insomnia; Suvorexant; Belsomra; Sleep disorder; Sleep
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders | interventions — suvorexant; Sugars

STUDY DESIGN:
Intervention Model Description: randomized cross-over trial of suvorexant and placebo for people with multiple sclerosis (MS), insomnia and fatigue
Who Masked: Participant, Investigator
Masking Description: investigator is blinded to randomization and results until study completion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Suvorexant (Experimental): Suvorexant - 10 mg (one tablet) taken by mouth once daily at bedtime with option to up-titrate to 20 mg (two tablets) taken by mouth once daily at bedtime.
  Interventions: Drug: Suvorexant
- Placebo (Placebo Comparator): Placebo - one tablet taken by mouth once daily at bedtime and two tablets taken by mouth daily at bedtime if subject up-titrates.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suvorexant — See detailed information in associated Arm Description.
  Other Names: Belsomra
  Arms: Suvorexant
Drug: Placebo — Sugar pill manufactured to mimic suvorexant 10 mg tablet.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
This study assesses the safety, tolerability, and efficacy of suvorexant in multiple sclerosis patients. Enrolled subjects will receive 2 weeks of treatment during treatment period 1 with either suvorexant or matching placebo (1:1). After treatment period 1, subjects will undergo a washout period of 1 week then 2 weeks of the alternate treatment (either suvorexant or placebo). The primary hypothesis is that suvorexant will provide greater improvement in sleep, as measured by symptom rating scales, compared to placebo.

DETAILED DESCRIPTION:
The target enrollment number is 30 people with multiple sclerosis who meet inclusion criteria. After informed consent is given, potential subjects will be screened to ensure they meet eligibility criteria. Subjects who meet eligibility criteria will complete baseline assessments and will then be randomized to receive 2 weeks of treatment (Treatment Period 1) with either suvorexant or matching placebo (1:1). The initial dose of suvorexant will be 10 mg at bedtime, with optional titration to 20 mg after 5-7 days. Study drug will be dispensed by an independent research pharmacist, keeping both study staff and the subject blinded. All subjects, whether in placebo or active arm, will receive a wearable sleep monitor to be worn for 7 days at baseline, and during both treatment periods. All subjects will keep 7-day sleep diaries at baseline and during each study period. At the end of Treatment Period 1 (2 weeks), subjects will undergo efficacy assessments with repeated clinical scales. Subjects will then go through a 1-week open-label off-drug washout period. Subjects will then be crossed over into the alternate treatment group, which will once again be double-blinded; those on active treatment (suvorexant) in Treatment Period 1 will be switched to placebo, and those on placebo in Treatment Period 1 will be switched to active treatment. Treatment Period 2 will also be 2 weeks long, and at the end of this, subjects will undergo final assessment with clinical scales.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis made at least 3 months prior based on McDonald criteria;
* Age 18-75 inclusive;
* Expanded Disability Status Scale (EDSS) 0- 7.5;
* Clinical stability defined as no multiple sclerosis exacerbation or change in disease modifying therapy for 60 days prior to screening;
* Screening Fatigue Severity Scale score of ≥4.0;
* Has Insomnia Disorder defined by diagnostic criteria published in the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5); namely, subject report of all of the following:

  * One of the following: difficulty initiating sleep; difficulty maintaining sleep; or early morning waking;
  * Sleep disturbance causes clinically significant distress or impairment in social, occupational, educational, academic, behavioral, or other important areas of functioning;
  * Sleep difficulty has occurred on 3 or more nights per week;
  * Sleep difficulty has been present for at least the past 3 months;
  * Sleep difficulty occurs despite adequate opportunity for sleep;
  * Insomnia is not explained by another sleep disorder;
  * Insomnia is not attributable to physiological effects of a consumed substance;
* May use other medications that could influence sleep, other than those specifically prohibited, as long as the dose is stable for 4 weeks preceding screening, with no dose changes during the study;
* Signed and dated Institutional Review Board-approved informed consent form before any protocol-specific screening procedures have been performed.

Exclusion Criteria:

* Use of potential multiple sclerosis-associated fatigue drugs within 3 days of screening until study completion, including modafinil, armodafinil, amantadine, methylphenidate, products with amphetamine or dextroamphetamine;
* Use of any of any prohibited medication (including Digoxin, benzodiazepines, barbiturates, opiates, Zolpidem, Zaleplon, Eszopiclone, moderate or strong CYP3A inhibitors, or strong inducers of CYP3A) from 3 days prior to screening to termination visit;
* Female who is breast-feeding, pregnant, or has the potential to become pregnant during the course of the study (fertile and unwilling/unable to use effective contraceptive measures);
* History of narcolepsy;
* Has a diagnosis of severe chronic obstructive pulmonary disease (COPD), defined by forced expiratory volume 1 (FEV1) < 50% of predicted on most recent available pulmonary function test (PFT). Pulmonary function test is not required if the subject has never been diagnosed with chronic obstructive pulmonary disease;
* Has a history of severe obstructive sleep apnea (OSA), with severe obstructive sleep apnea defined as having an apnea-hypopnea index (AHI) > 30 on prior polysomnograph (PSG). Polysomnograph is not required if there is no history of obstructive sleep apnea;
* Is concurrently using other central nervous system (CNS) depressants, including alcohol, except that one alcoholic drink per day will be allowed for those with normal hepatic function provided the drink is consumed at least 2 hours prior to or 8 hours after taking the study drug. Medical marijuana is allowed if consumed at the patient's usual dose at least 2 hours prior to or 8 hours after taking the study drug. Recreational marijuana is not allowed from screening until end of study;
* Has evidence at screening of severe hepatic impairment as defined by a Child-Pugh score > 10;
* Cognitive impairment that in the opinion of the investigator would prevent completion of study procedures or the ability to provide informed consent;
* Suicidality or severe depression as measured by screening Beck Depression Inventory II (BDI) score > 28 or score of >1 on Beck Depression Inventory II Question 9 (suicidality screen) at any time during the study;
* Any other serious and/or unstable medical condition.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore R Brown, MD, MPH, Principal Investigator — EvergreenHealth Multiple Sclerosis Center
Locations (1):
- EvergreenHealth Multiple Sclerosis Center, Kirkland, Washington, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 36 subjects were enrolled
Pre-assignment Details: Subjects were randomized 1:1 to Suvorexant - 10 mg (one tablet) taken by mouth once daily at bedtime with option to up-titrate to 20 mg (two tablets) taken by mouth once daily at bedtime or matching placebo. The subjects crossed over to opposite treatment for two weeks following a 1-week washout
Groups:
- Suvorexant Followed by Placebo: Suvorexant - 10 mg (one tablet) taken by mouth once daily at bedtime with option to up-titrate to 20 mg (two tablets) taken by mouth once daily at bedtime.
  Suvorexant: See detailed information in associated Arm Description.
- Placebo Followed by Suvorexant: Placebo - one tablet taken by mouth once daily at bedtime and two tablets taken by mouth daily at bedtime if subject up-titrates.
  Placebo: Sugar pill manufactured to mimic suvorexant 10 mg tablet.
Period: Overall Study
Arm/Group | Suvorexant Followed by Placebo | Placebo Followed by Suvorexant
Started (Crossover trial, all subjects received both treatments) | 18 (crossover trial. All subjects received both treatments) | 18
Completed (1) | 17 | 18
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Suvorexant Followed by Placebo: Suvorexant - 10 mg (one tablet) taken by mouth once daily at bedtime with option to up-titrate to 20 mg (two tablets) taken by mouth once daily at bedtime. After one week washout, Placebo - one tablet taken by mouth once daily at bedtime and two tablets taken by mouth daily at bedtime if subject up-titrates.
  Suvorexant: See detailed information in associated Arm Description. Placebo: Sugar pill manufactured to mimic suvorexant 10 mg tablet.
- Placebo Followed by Suvorexant: Placebo - one tablet taken by mouth once daily at bedtime and two tablets taken by mouth daily at bedtime if subject up-titrates. After one week washout, Suvorexant - 10 mg (one tablet) taken by mouth once daily at bedtime with option to up-titrate to 20 mg (two tablets) taken by mouth once daily at bedtime.
  Suvorexant: See detailed information in associated Arm Description. Placebo: Sugar pill manufactured to mimic suvorexant 10 mg tablet.
- Total: Total of all reporting groups
Arm/Group | Suvorexant Followed by Placebo | Placebo Followed by Suvorexant | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.333 (13.412) | 55.118 (10.775) | 52.657 (12.616)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 17 | 18 | 35
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Northwest United States of America
  participants
    United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change in Insomnia Severity Index (ISI) Score
Description: 7-question survey assessing symptoms of insomnia over the past week. Maximum score is 28, minimum is 0, with higher scores indicating greater severity.
  Guidelines for Scoring/Interpretation:
  Add scores for all seven items = _____ Total score ranges from 0-28 0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate
Time Frame: Change from Baseline to 2 Weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 35 | 35
score on a scale | -4 [-8 to -2] | -2 [-5 to 0]

2. Secondary Outcome: Change in Modified Fatigue Index Scale (MFIS) Score
Description: This scale has 21 items with physical, cognitive and psychosocial questions regarding their fatigue levels. Subjects will complete the Modified Fatigue Index Scale (MFIS) as the first test conducted on the day of visit. Their ratings on the 21-item questionnaire will be based on their fatigue experience over the previous 1 week. Each question is on a scale from 0 to 4. Higher scores represent worse fatigue. Minimum score is 0 and maximum score is 84.
Time Frame: Change from Baseline to 2 Weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 35 | 35
score on a scale | -10.5 [-16.5 to -3.5] | -8.5 [-15 to 1.5]

3. Secondary Outcome: Patient Global Impression of Change
Description: This is a single question: "How would you rate change in your level of physical and mental function, during the study?" Responses range from "Extremely improved", "Much improved", "Slightly improved", "No change", "Slightly worse", "Much worse", and "Extremely worse". Higher score indicates improvement. Scale is 0-5 given responses. 0 is minimum, 5 is maximum.
Time Frame: Change from Baseline to 2 Weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 35 | 35
score on a scale | 0 [0 to 1] | 0 [0 to 1]

4. Secondary Outcome: Fatigue Visual Analog Scale
Description: 0-100 scale rating fatigue with 0 being not fatigued at all, 100 being fatigue as bad as can be. Patients are instructed to place an "X" on the scale based on their overall level of fatigue. On the low-end of the scale are feelings of being awake and alert, having high-energy and vigor. On the high end of the scale are feelings of tiredness, drowsiness, sluggishness, low-energy, lassitude.
Time Frame: Change from Baseline to 2 Weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 35 | 35
score on a scale | -5 [-20 to 5.61] | -5 [-15 to 0]

5. Other Pre Specified Outcome: Sleep Latency
Description: A measure of minutes between being awake and falling asleep.
Time Frame: Change from Baseline to 2 Weeks
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 35 | 35
Minutes | -4.29 [-26.05 to 5.61] | -2.8 [-17.45 to 10.38]

6. Other Pre Specified Outcome: Subjective Quality of Sleep (sQUAL)
Description: This is a single question, "How would you describe the quality of your sleep last night?" There are 4 choices to answer: 1= poor, 2 = fair, 3= good, 4= excellent. 1 is Minimum, 4 is maximum. A higher score means a better outcome.
Time Frame: Change from Baseline to 2 Weeks
Measure: Median (Inter-Quartile Range); unit: Score on a Scale
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 35 | 35
Score on a Scale | 0 [0 to 1] | 0 [0 to 1]

ADVERSE EVENTS:
Time Frame: 5 weeks from Baseline to end of study.
Description: All adverse events were captured after the subject baseline date when they were randomized into either arm. For each reported adverse event, the subjects were followed until resolution of the adverse event or the end of the study.
Arm/Group | Suvorexant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 7/35 | 1/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suvorexant (N=35) | Placebo (N=35)
Headache (General disorders) | 3 (3) | 1 (1)
Sleep Disturbance (General disorders) | 2 (2) | 0 (0)
Dry Mouth (General disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Increased Depression (Psychiatric disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This was a small study done at two centers with treatment windows limited to two weeks including dose escalation. A two-week exposure may have been inadequate to elicit full treatment effect. It is also possible that the one-week washout period was insufficient.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT03110315/Prot_SAP_000.pdf